CLINICAL TRIAL: NCT07306078
Title: Attentional Ability and Resilience to Alcohol Use Disorder: Neurocognitive Mechanisms: Protocol Two
Brief Title: Methylphenidate and Response to Alcohol Cues
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB202500591; R01AA032400 (NIH)
Record Dates: First submitted 2025-12-03; First posted 2025-12-29 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-04

CONDITIONS: Alcohol Use Disorder
Keywords: fMRI; methylphenidate; ritalin; attention; alcohol
MeSH Terms: conditions — Alcoholism | interventions — Methylphenidate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Crossover 1: methylphenidate, placebo (Experimental): methylphenidate (single dose, oral, 20 mg, immediate release) followed by placebo (single dose, oral)
  Interventions: Drug: Methylphenidate Pill; Other: Placebo Pill
- Crossover 2: placebo, methylphenidate (Experimental): placebo (single dose, oral) followed by methylphenidate (single dose, oral, 20 mg, immediate release)
  Interventions: Drug: Methylphenidate Pill; Other: Placebo Pill

INTERVENTIONS:
Drug: Methylphenidate Pill — Encapsulated methylphenidate
Other: Placebo Pill — Encapsulated placebo

SUMMARY:
The purpose of this study is to determine whether changes in attention levels related to taking a single dose of a medication called methylphenidate, also known as Ritalin, affects responses to alcohol cues. The study will observe the effects of methylphenidate or a placebo on neural and craving responses to alcohol cues through fMRI and behavioral testing. Participants will be involved in one remote and two in-person sessions.

DETAILED DESCRIPTION:
Recent studies have revealed a robust link between attentional ability and resilience against stress-related psychopathology, in general, and against alcohol use disorder (AUD) specifically. For example, self-reported attentional ability correlates with scales of psychological resilience and with lower alcohol misuse in at-risk individuals. One mechanism by which attention may relate to resilience in AUD is through its effects on alcohol cue reactivity. Exposure to alcohol cues can induce motivation to drink alcohol for those with AUD. Leveraging the high rates of co-morbidity of AUD and attention-deficit/hyperactivity disorder, this pilot study seeks to demonstrate whether experimentally enhancing attention in individuals with alcohol misuse reduces markers of addiction severity (i.e., craving and attentional bias responses to alcohol cues) and will explore the neural and behavioral mechanisms. Methylphenidate not only improves sustained attention, but in users of cocaine and methamphetamine, it was previously shown to reduce craving, attentional bias, and neural responses to viewing drug-related cues. This study will use this commonly-prescribed medication as a pharmacological probe of attentional processes related to alcohol use disorder. It is hypothesized that acute methylphenidate-associated attentional enhancement will engage compensatory brain mechanisms that will lead to attenuated craving, reduced attentional bias, and modulated neural responses to alcohol cues in young adults. Fifty young adults reporting hazardous alcohol use will be recruited for a double-blind, placebo-controlled, within-subjects experiment to test the effects of an acute 20 mg methylphenidate administration to increase attention on cue-induced alcohol craving [during functional magnetic resonance imaging (fMRI)] and attentional bias. Subjects will also perform computerized tasks of general attention with non-alcohol-related stimuli.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-25 years
* Meets DSM-5 criteria for Alcohol Use Disorder -OR- score on the Alcohol Use Disorders Identification Test (AUDIT) of >=8
* Fluent in English
* Normal or corrected to normal vision

Exclusion Criteria:

* Meets DSM-5 criteria for psychotic disorders, neurological disorders, or substance use disorders other than Alcohol Use Disorder.
* Participant routinely uses psychoactive drugs or medications except for non-dependent marijuana or nicotine use (due to common use of these substances in individuals with Alcohol Use Disorder).
* Participant has contraindications for taking methylphenidate.
* Participant has contraindications for being in an MRI machine
* Self-reported history of high blood pressure over 140/90 or consistent readings of 140/90 or above upon arrival for a session.
* History of seizure disorder
* Liver disease
* Participant is currently pregnant or trying to become pregnant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Neural responses to cues | 15 minutes
  Whole-brain cue-elicited fMRI responses will be examined by contrasting activation following alcohol images with brain activation following neutral images. Regions-of-interest analysis will focus on anterior cingulate cortex, dorsal striatum, ventral striatum, and amygdala.

SECONDARY OUTCOMES:
Self-reported craving | 15 minutes
  Craving following presentation of alcohol and neutral images will be reported using 0-10 visual analog scales. Differences in craving following the alcohol images and craving following the neutral images will be tested.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
The final dataset will include brain imaging, behavioral, and self-report data obtained from task (viewing of alcohol pictorial cues), self-ratings of craving during the task scan, computerized tasks of attention, and interview and survey measures of mental health and substance use. De-identified individual-participant level (IPD) raw data will be shared. Appropriate measures such as de-facing T1 anatomical MRI images using software for this purpose (e.g., mri_deface) will be used for data de-identification prior to sharing, and informed consent forms will reflect those plans.
Supporting Information: CSR
Time Frame: 2028-2033
Access Criteria: Scientists with access to the NIH-managed data repository will have access to the IPD.